CLINICAL TRIAL: NCT00646334
Title: A Randomised, Multi-center, Prospective, Observer and Patient Blind Study to Evaluate AESCULAP Optilene® Mesh Elastic Versus Ethicon Ultrapro® Mesh in Incisional Hernia Repair
Brief Title: Comparative Study of AESCULAP Optilene® Mesh Elastic Versus Ethicon Ultrapro® Mesh in Incisional Hernia Repair
Acronym: Optilene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAG-G-H-0505
Record Dates: First submitted 2008-03-18; First posted 2008-03-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Incisional Hernia Repair
Keywords: Large Pore Size Propylene Mesh; Incisional Hernia; Randomized Controlled Double-blind Study
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Optilene® Mesh Elastic
  Interventions: Device: Mesh Implantation
- B (Active Comparator): Ultrapro® Mesh
  Interventions: Device: Mesh Implantation

INTERVENTIONS:
Device: Mesh Implantation — An elective incisional Hernia repair is performed by using Optilene® Mesh Elastic, a lightweight and large pore mesh, knitted from monofilament polypropylene. Due to the multidirectional elasticity the mesh is able to adapt to all movements taking place in the abdominal wall.
  Other Names: Optilene® Mesh Elastic
  Arms: A
Device: Mesh Implantation — Ultrapro® Mesh is a knitted, partly absorbable, lightweight mesh, consisting of equal parts of nonabsorbable polypropylene and absorbable polyglecaprone (Monocryl®). Polyglecaprone is fully absorbed in the body by hydrolysis. The addition of polyglecapron filament is only intended to reinforce the mesh to allow a convenient intraoperative handling and mesh placement, without additional function. Ultrapro® is an elastic mesh having enlarged elasticity cross to the blue strips.
  Other Names: Ultrapro® Mesh
  Arms: B

SUMMARY:
Optilene® Mesh Elastic and Ultrapro® Mesh will be used for incisional hernia repair. The primary objective of this clinical study is to demonstrate that Optilene® Mesh Elastic is superior to Ultrapro® Mesh in incisional hernia repair in matter of the physical function score from the SF-36 questionnaire 21 days after mesh insertion. Secondary objectives include the patient's daily activity, the rating of patients pain and the wound assessment determined on several occasions during the six months observation time.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients >=18 years
* Female patients are incapable of pragnancy or must be using adequate contraception and are not in lactation
* Patients wiht vertical aponeurotic incisions only
* Incisional hernia with hernia size >= 3 cm
* Patient is capable to understand and to follow the instructions
* written informed consent
* no mesh implantation at the same site during a previous operation
* immune competence of patient

Exclusion Criteria:

* Simultanous participation in an investigational drug or medical device study
* Patients < 18 years old
* Incisional Hernia withe a hernia size < 3 cm
* Repair of an acute incarcerated hernia
* Previous mesh repair at the same site
* Patient with other than vertical aponeurotic incisions
* Enterotomy to be performed during hernia repair at Surgery
* Patient is on anti-coagulations-therapy
* Patient is known or assessed to be non-compliant
* Additional surgical treatment at the same time (e.g. cholecystectomy)
* Immune incompetence of patient (e.g. chemotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Physical function score of the SF-36 questionnaire | 21 days after insertion

SECONDARY OUTCOMES:
physical function score from the SF-36 questionnaire | 6 months postoperatively
patient's daily activity | 6 months postoperatively
patient's pain | 6 months postoperatively
wound assessment | 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kuthe, Dr., Principal Investigator — DRK Krankenhaus Clementinenhaus, Hannover; Rainer Engemann, Prof. Dr., Principal Investigator — Klinikum Aschaffenburg, Chirurgische Klinik; Jens Kuhlgatz, Dr., Principal Investigator — Albert-Schweitzer-Krankenhaus, Klinik fuer Allgemein- und Viszeralchirurgie, Zentrum fuer Minimalinvasive Chirurgie, Northeim; Peter Kienle, Prof. Dr., Principal Investigator — Universitaetsklinikum Mannheim, Chirurgische Klinik; Markus Buechler, Prof.Dr.Dr., Principal Investigator — Universitaetsklinikum Heidelberg, Abt. fuer Allgemein-, Viszeral-, Unfallchirurgie und Poliklinik; Moritz von Frankenberg, Dr., Principal Investigator — Krankenhaus Salem, Chirurgische Abteilung, Heidelberg
Locations (6):
- Germany (6):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Krankenhaus Salem, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Mannheim, Mannheim, Baden-Wurttemberg
  - Klinikum Aschaffenburg, Aschaffenburg, Bavaria
  - Andreas Kuthe, Hanover, Lower Saxony
  - Albert-Schweitzer Krankenhaus, Northeim, Lower Saxony

REFERENCES:
- [Background] Cassar K, Munro A. Surgical treatment of incisional hernia. Br J Surg. 2002 May;89(5):534-45. doi: 10.1046/j.1365-2168.2002.02083.x. PMID 11972542
- [Background] Schumpelick V, Arlt G, Klinge U. [Versorgung von Nabelhernien und Narbenhernien]. Dt. Aerzteblatt 94, Heft 51-52. Dez. 1997 (35)
- [Background] Klinge U, Conze J, Limberg W, Brucker C, Ottinger AP, Schumpelick V. [Pathophysiology of the abdominal wall]. Chirurg. 1996 Mar;67(3):229-33. German. PMID 8681695
- [Background] Klinge U, Conze J, Klosterhalfen B, Limberg W, Obolenski B, Ottinger AP, Schumpelick V. [Changes in abdominal wall mechanics after mesh implantation. Experimental changes in mesh stability]. Langenbecks Arch Chir. 1996;381(6):323-32. doi: 10.1007/BF00191312. German. PMID 9082105
- [Background] Schumpelick V, Lloyd M. Meshes: benefits and risks, 9 Polypropylene: The standard of Mesh Materials. Nyhus Editors, Springer Verlag, 2004: 101-103
- [Background] Beets GL, Go PM, van Mameren H. Foreign body reactions to monofilament and braided polypropylene mesh used as preperitoneal implants in pigs. Eur J Surg. 1996 Oct;162(10):823-5. PMID 8934114
- [Background] Klinge U, Klosterhalfen B, Birkenhauer V, Junge K, Conze J, Schumpelick V. Impact of polymer pore size on the interface scar formation in a rat model. J Surg Res. 2002 Apr;103(2):208-14. doi: 10.1006/jsre.2002.6358. PMID 11922736
- [Background] Benhidjeb T, Baerlehner E, Anders S. Laparoskopische Narbenhernien Reparation: Muss das Netz fuer die Intraperitoneale Onlay-Mesh-Technik besondere Eigenschaften haben?; Chir. Gastroenterol. 2003; 19(Suppl.2): 16-22
- [Background] Rosen HR, Gyasi A; Retromuskulaere Kunststoffnetzimplantation von Narbenhernien; Chir. Gastroenterol.; 2003; 19 (Suppl. 2); 39-45
- [Background] Rosch R, Junge K, Stumpf M, Klinge U, Schumpelick V, Klosterhalfen B; Welche Anforderungen sollte ein ideales Netz erfuellen?; Chir. Gastroenterol.; 2003; 19 (Suppl. 2); 7-11
- [Background] Schumpelick V, van Ackeren H, Klinge U; Hernien; Thieme Verlag, 2000; 266-267
- [Background] Seiler C, Baumann P, Kienle P, Kuthe A, Kuhlgatz J, Engemann R, V Frankenberg M, Knaebel HP. A randomised, multi-centre, prospective, double blind pilot-study to evaluate safety and efficacy of the non-absorbable Optilene Mesh Elastic versus the partly absorbable Ultrapro Mesh for incisional hernia repair. BMC Surg. 2010 Jul 12;10:21. doi: 10.1186/1471-2482-10-21. PMID 20624273
- [Result] Rickert A, Kienle P, Kuthe A, Baumann P, Engemann R, Kuhlgatz J, von Frankenberg M, Knaebel HP, Buchler MW. A randomised, multi-centre, prospective, observer and patient blind study to evaluate a non-absorbable polypropylene mesh vs. a partly absorbable mesh in incisional hernia repair. Langenbecks Arch Surg. 2012 Dec;397(8):1225-34. doi: 10.1007/s00423-012-1009-6. Epub 2012 Oct 3. PMID 23053458